CLINICAL TRIAL: NCT04846452
Title: Sintilimab Combined With Anlotinib Hydrochloride and Standard Platinum-Containing Dual-Agent Chemotherapy in Non-Small Cell Lung Cancer (NSCLC) as First-Line Treatment: A Single-Arm, Prospective and Exploratory Clinical Study
Brief Title: Sintilimab, Anlotinib Hydrochloride and Platinum-Containing Dual-Agent Chemotherapy in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SR-088
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Metastatic NSCLC; Recurrent NSCLC; Advanced Non-Small Cell Squamous Lung Cancer
Keywords: Metastatic NSCLC; Recurrent NSCLC; Advanced NSCLC; Sintilimab; Anlotinib Hydrochloride; Chemotherapy; First-Line Treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; anlotinib; Pemetrexed; Cisplatin; Carboplatin; Combined Modality Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSCLC patients with negative driver genes (Experimental): Patients with negative driver genes advanced or metastatic NSCLC will receive sintilimab combined with anlotinib hydrochloride and platinum-containing dual-agent chemotherapy regimens as first-line treatment.
  Interventions: Drug: Sintilimab + Anlotinib + Pemetrexed + Cisplatin or Carboplatin; Drug: Sintilimab + Anlotinib + Albumin Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: Sintilimab + Anlotinib + Pemetrexed + Cisplatin or Carboplatin — Patients with non-squamous NSCLC will receive sintilimab, anlotinib hydrochloride, pemetrexed, and cisplatin or carboplatin.
  Other Names: combination therapy
Drug: Sintilimab + Anlotinib + Albumin Paclitaxel + Carboplatin — Patients with squamous NSCLC will receive sintilimab, anlotinib hydrochloride, albumin paclitaxel, and carboplatin.
  Other Names: combination therapy

SUMMARY:
This is a single-arm, prospective, exploratory clinical study aiming to evaluate the efficacy and safety profile of sintilimab combined with anlotinib hydrochloride and platinum-containing dual-agent chemotherapy regimens in advanced or metastatic NSCLC as first-line treatment. Totally 40 patients with negative driver genes (20 patients of squamous cell carcinoma, 20 patients of non-squamous cell carcinoma) are to be enrolled.

DETAILED DESCRIPTION:
Sintilimab (200 mg intravenously, once every 3 weeks; Cinda Bio-Suzhou Co., Ltd., Suzhou, Jiangsu, China) and anlotinib hydrochloride (12 mg orally, once daily before breakfast; CTTQ, Lianyungang, Jiangsu, China) are to be administered as first-line therapy in NSCLC. Besides, patients with non-squamous NSCLC will also receive pemetrexed and cisplatin or carboplatin. Meanwhile, patients with squamous NSCLC will also receive albumin paclitaxel and carboplatin. Patients assessing as CR/PR/SD will continue to receive a maintenance treatment after 4-6 cycles of treatment. Patients with non-squamous NSCLC will be treated with sintilimab + anlotinib hydrochloride + pemetrexed chemotherapy regimen while patients with squamous NSCLC will be treated with sintilimab + anlotinib hydrochloride to maintain treatment for 2 years until disease progression, intolerable toxicity, death, and patient request for discontinuation or starting new anti-tumor treatment.

Observations and assessments will be conducted before treatment, on day 7, 21 of cycle 1, on day 21 of cycle 2, every 2 cycles (42 days) during the following cycles, and after treatment. Follow-up for survival status and subsequent antineoplastic therapy data collecting will be performed by telephone interview or face-to-face every 6 weeks after treatment until disease progression, death, or end of the study (whichever occurs first).

This study will be divided into two stages: the safety lead-in period and the preliminary efficacy evaluation period. The first stage is the safety lead-in period. 3 patients with squamous NSCLC and 3 patients with non-squamous NSCLC will be enrolled to evaluate the combined therapy safety. The first 6 patients will continue to be observed from the beginning of the combined treatment until the 6th patient has been treated for 2 cycles (6 weeks). If there are less than or equal to 2 patients with intolerable side effects, they will enter the next stage. A total of 40 patients (20 patients with squamous NSCLC, 20 patients of non-squamous NSCLC) will be enrolled, and the safety and efficacy of the combined treatment will be initially evaluated. All statistics will be analyzed by statistical analysis software (SAS) 9.2 (or higher version). The single-sided 0.05 superiority hypothesis test will be used to test statistics and the comparison between groups will give a 95% confidence interval and p-value.

Efficacy is to be analyzed in the full analysis set (FAS), the response evaluable set (RES), and the per-protocol set (PPS). Safety is to be analyzed in safety set (SS) including all assigned patients who receive at least one dose of study combined therapy and have safety records of medication. Statistical descriptions of subject distribution, demographic data, and baseline characteristics will be performed. For study endpoints, the Kaplan-Meier method is to be applied for the PFS and OS curve with estimation for median PFS, median OS, and 95% CI. ORR= (CR+PR) / sample size×100%; DCR= (CR+PR+SD) / sample size×100%. The 95% CI of the ORR and DCR is to be calculated by an exact binomial method based on the F distribution. For safety analysis, only treatment-emergent adverse events (TEAE) will be included and analyzed in this experiment, which is defined as AEs that are post-dose or heavier than the baseline. Medical Dictionary for Regulatory Activities (MedDRA), system organ class (SOC), preferred terms (PT) and NCI CTCAE 5.0 will be used to standardize and classify all adverse events and summarize the incidence of AEs and association with treatments.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntary provision of informed consent.
* 2. Males or females aged 18-75.
* 3. Histological or cytologically confirmed NSCLC, metastatic or recurrent (stage IV), non-resectable or radical radio-chemotherapy locally advanced (stage IIIB-IIIC).
* 4. Not suitable for targeted therapy (patients with non-squamous NSCLC have no EGFR, ALK, or ROS1 gene mutation)
* 5. At least one lesion can be measured by imaging.
* 6. Have not received systemic treatment in the past.
* 7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
* 8. Life expectancy ≥ 3 months.
* 9. Female of childbearing age must have a negative pregnancy test (serum or urine) within 7 days before enrolment.

Exclusion Criteria:

* 1. Histological or cytologically confirmed small cell lung cancer (SCLC), including lung cancer mixed with SCLC and NSCLC.
* 2. Received radiation therapy within 6 weeks.
* 3. Diagnosed with other malignant diseases other than NSCLC within 5 years.
* 4. Have participated in other interventional clinical research treatments now or within 4 weeks.
* 5. Have previously received targeted therapy.
* 6. Received Chinese patent medicines with anti-lung cancer indications or immunomodulatory drugs within 2 weeks.
* 7. Have active autoimmune diseases requiring systemic treatment within 2 years.
* 8. Received systemic glucocorticoid therapy or immunosuppressive therapy within 7 days.
* 9. Clinically uncontrollable pleural effusion/abdominal effusion.
* 10. Known allogeneic organ transplantation or hematopoietic stem cell transplantation.
* 11. Known to be allergic to study drug.
* 12. Have been vaccinated with the live vaccine within 30 days.
* 13. Pregnant or breastfeeding females.
* 14. Other serious hazards to the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Object response rate (ORR) | Time Frame: Up to 24 moths.
  Containing the incidence of complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months.
  From allocation to first disease progression confirmed by imaging modalities or all cause death, whichever occurs first.
Disease control rate (DCR) | Up to 24 months.
  Containing the incidence of complete response (CR), partial response (PR) and stable disease (SD).
Duration of Remission (DOR) | Up to 24 months.
  The time interval from disease remission to disease progression or death (whichever occurs first).
Overall survival (OS) | Up to 24 months.
  From allocation to any cause death or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lingxiang Liu, Physician, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD and all IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.
Access Criteria: IPD will be shared with other related clinical trials or systematic reviews after reviewing requests by the chief investigator and examiners.

REFERENCES:
- [Background] McDermott DF, Atkins MB. PD-1 as a potential target in cancer therapy. Cancer Med. 2013 Oct;2(5):662-73. doi: 10.1002/cam4.106. Epub 2013 Jul 21. PMID 24403232
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Travis WD, Brambilla E, Nicholson AG, Yatabe Y, Austin JHM, Beasley MB, Chirieac LR, Dacic S, Duhig E, Flieder DB, Geisinger K, Hirsch FR, Ishikawa Y, Kerr KM, Noguchi M, Pelosi G, Powell CA, Tsao MS, Wistuba I; WHO Panel. The 2015 World Health Organization Classification of Lung Tumors: Impact of Genetic, Clinical and Radiologic Advances Since the 2004 Classification. J Thorac Oncol. 2015 Sep;10(9):1243-1260. doi: 10.1097/JTO.0000000000000630. PMID 26291008
- [Result] Barbee MS, Ogunniyi A, Horvat TZ, Dang TO. Current status and future directions of the immune checkpoint inhibitors ipilimumab, pembrolizumab, and nivolumab in oncology. Ann Pharmacother. 2015 Aug;49(8):907-37. doi: 10.1177/1060028015586218. Epub 2015 May 19. PMID 25991832
- [Result] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Result] Jiang S, Liang H, Liu Z, Zhao S, Liu J, Xie Z, Wang W, Zhang Y, Han B, He J, Liang W. The Impact of Anlotinib on Brain Metastases of Non-Small Cell Lung Cancer: Post Hoc Analysis of a Phase III Randomized Control Trial (ALTER0303). Oncologist. 2020 May;25(5):e870-e874. doi: 10.1634/theoncologist.2019-0838. Epub 2020 Feb 20. PMID 32077550